CLINICAL TRIAL: NCT06498141
Title: MucinB5 rs (35705950) Gene Polymorphism and Leucocytes Telomere Length in Relation to Interstitial Lung Diseases.
Brief Title: MucinB5 Gene Polymorphism and Leucocytes Telomere Length in Interstitial Lung Diseases
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Amera Morad Foad, Assistant Professor of Medical Biochemistry, Sohag University
Other Study IDs: Soh-Med-23-02-21
Record Dates: First submitted 2024-07-06; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Mucin B5 rs (35705950) Gene Polymorphism in Interstitial Lung Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diseased: patients with interstitial lung diseases fulfilling the inclusion criteria.
- Control: Healthy subjects

SUMMARY:
This is an observertional study aimed at Study the association between Mucin B5 rs (35705950) gene polymorphism and Leucocytes telomere length in relation to interstitial lung diseases.

ELIGIBILITY:
Inclusion Criteria:

This study will include patients with interstitial lung diseases aged above 18 years old.

Exclusion Criteria:

* patients with emphysema or obstructive lung diseases.
* patients with active cancer
* End stage renal failure (GFR < 30 ml/min) or on dialysis
* Liver cell failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with interstitial lung diseases in our center in sohag university hospital
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
MucinB5 rs (35705950) gene polymorphism | 6 Months
  whether homogenetic or heterogenetic
Leucocytes telomere length | 6 months
  Measurement of the relative length of WBCs telomere in patints with interstitial pulmonary fibrosis

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university hosoital, Sohag, Egypt